CLINICAL TRIAL: NCT05585840
Title: The Effect of Biofeedback-Based Virtual Reality Game on Pain, Fear and Anxiety Levels During Insertion of Port Needle in Children
Brief Title: The Effect of Biofeedback-Based Virtual Reality Game on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching and Research Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Eysan Hanzade Umac
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Cancer
Keywords: port catheter; pediatric oncology; pain; anxiety; fear; biofeedback; virtual reality
MeSH Terms: conditions — Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback-based virtual reality group/Intervention (Experimental): When approaching the moment of the procedure (2 minutes before), children will be asked to put on the virtual reality glasses, saturation probe and respiratory sensor in addition to routine care. At this stage, the child will be assisted by the researcher. The launch of the mobile application on the researcher's phone will be provided just before the port needle placement (1 minute before). In this process, the child will provide biofeedback to the game with regular and deep breathing behavior. The game will end when the port pin placement is complete.
  Interventions: Device: Biofeedback-based virtual reality game
- Control group (No Intervention): In the pediatric oncology unit where the study will conduct, there is no standard pharmacological and non-pharmacological application use to reduce pain, anxiety, and fear during intervention. Family presence and positive encouragement are used in routine care. For children in this group, port catheter needle insertion will be performed in accordance with their clinical routines.

INTERVENTIONS:
Device: Biofeedback-based virtual reality game — The application will be a biofeedback-based virtual reality game developed by the researchers in collaboration with engineering in line with the literature review.
  Arms: Biofeedback-based virtual reality group/Intervention

SUMMARY:
The needles of port catheters, which are often used in childhood cancer treatment, must be changed every 5-7 days, which causes pain, anxiety, and fear in children every 5-7 days In recent years, the usage of virtual reality has grown to distract children during port catheter needle insertion. But it's not always easy for children to switch their attention to something else. A good child distractor must be sensory-stimulating, developmentally appropriate, and highly interactive.

DETAILED DESCRIPTION:
Today, virtual reality applications have advanced, and software that provides biofeedback with breathing has improved engagement with the user. Our aim in this study is to examine the effect of biofeedback-based virtual reality games on pair, fear and anxiety levels during insertion of port needle insertion in children.

The randomized control trial design will be used, and The CONSORT list will be used to guide the research. This study will be conducted at the 62 pediatric oncology patients (31 experiment/ 31 control) aged 6-12 years. This study will be carry out in a university hospital in Istanbul, Turkey between January 2023, and June 2023. The research data will collect from the children's self-reports and parents through a survey form and scales. Children's pain will evaluate by the children and parent with Wong-Baker Faces Pain Rating Scale, child fear will evaluate by the children and parent with 'Child Fear Inventory', and child anxiety will evaluate by the children and parent with 'Child Anxiety Statement Scale'.

ELIGIBILITY:
Inclusion criteria:

* Between the ages of 6-12,
* Requires venous access
* Diagnosed with childhood cancer,
* Volunteers with at least one venous access experience.

Exclusion Criteria:

* With neurodevelopmental delay,
* Difficulty in verbal communication
* Auditory or visual impairment
* Those who have used analgesics in the last 24 hours and have a history of needle phobia.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale | Evaluation will be done approximately 5 minutes after port catheter needle placement.
  Wong-Baker Faces Pain Rating Scale. It is used in the assessment of pain in children. The scale consists of six facial expressions. Facial expressions range from 0 points of "no pain-very happy" to 10 points of "unbearable pain-crying". It is commonly used in children aged 3-18. It has good validity and reliability for the measurement of pain severity and is psychometrically suitable and widely used in clinical practice.
The Child Fear Scale (CFS) | It will be evaluated 5-minute before the insertion of port needle.
  The Child Fear Scale (CFS). It measures procedure-related fear in children. It consists of five sex-neutral faces; 0 (no fear) - 4 (extreme fear). It is based on the Faces Anxiety Scale. The FAS changed developmentally to the CFS. It can be used by the parents during the procedure for 5-10 years old children. Assessment of construct validity revealed high concurrent convergent validity with another self-report measure of fear and moderate discriminant validity with coping and distress behavior.
The Child Fear Scale (CFS) | It will be evaluated 5-minute after the insertion of port needle.
  The Child Fear Scale (CFS). It measures procedure-related fear in children. It consists of five sex-neutral faces; 0 (no fear) - 4 (extreme fear). It is based on the Faces Anxiety Scale. The FAS changed developmentally to the CFS. It can be used by the parents during the procedure for 5-10 years old children. Assessment of construct validity revealed high concurrent convergent validity with another self-report measure of fear and moderate discriminant validity with coping and distress behavior.
The Children's Anxiety Meter (CAM) | It will be evaluated 5-minute before the insertion of port needle.
  The Children's Anxiety Meter (CAM). It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.CAM were administered by the researcher to the children to assess their anxiety levels about blood draw before and after the blood draw procedure.
The Children's Anxiety Meter (CAM) | It will be evaluated 5-minute after the insertion of port needle.
  The Children's Anxiety Meter (CAM). It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.CAM were administered by the researcher to the children to assess their anxiety levels about blood draw before and after the blood draw procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Hanzade Umaç, Study Director — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No